CLINICAL TRIAL: NCT07383844
Title: Analysis of Barriers and Facilitators to Adapted Physical Activity for Pediatric Patients With Chronic Inflammatory Bowel Diseases
Acronym: Feels-Mici
Status: Recruiting | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 25-HPNCL-08 Feels-MICI; 2025-A02019-40 (Other: id-rcb)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease (Crohn's Disease; Ulcerative Colitis)
Keywords: physical activity
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric IBD participants (questionnaires + interview): This study does not involve any therapeutic or behavioral intervention. The "intervention" corresponds to data collection during a single visit: participants complete two self-administered questionnaires (CAPAS-Q and IMPACT-III) and participate in a semi-structured interview about perceived barriers and facilitators to physical activity. No counseling, training, or treatment is provided.
  Interventions: Other: IMPACT-III questionnaires; Other: Data collection: CAPAS-Q; Other: semi-structured interview

INTERVENTIONS:
Other: IMPACT-III questionnaires — Participants complete the self-administered questionnaires IMPACT-III)
Other: Data collection: CAPAS-Q — Participants complete the self-administered questionnaires CAPAS-Q.
Other: semi-structured interview — participate in a semi-structured interview about perceived barriers and facilitators to physical activity. No counseling, training, or treatment is provided.

SUMMARY:
This study aims to identify perceived barriers and facilitators to regular physical activity among children and adolescents with inflammatory bowel disease (IBD) followed in pediatric gastroenterology. Approximately 60 participants aged 10-17 years will complete two self-administered questionnaires (CAPAS-Q for physical activity/sedentary behavior and IMPACT-III for health-related quality of life) and take part in a single semi-structured interview exploring experiences, obstacles, and levers to support sustainable physical activity. Relevant clinical data (disease characteristics, treatment and selected routine clinical parameters) will be extracted from the medical record. Participation is limited to one visit (about 45-60 minutes) during a routine hospital appointment, with no additional intervention or follow-up required.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 to 17 years at inclusion.
* Diagnosed inflammatory bowel disease (Crohn's disease or ulcerative colitis) confirmed and diagnosed for at least 6 months.
* Followed in the pediatric gastroenterology department at Hôpital Lenval (CHU de Nice).
* Sufficient cognitive and language abilities to understand questionnaires and participate in an individual interview.
* Affiliated to, or beneficiary of, a social security scheme.
* no parental objection to participation (non-opposition).

Exclusion Criteria:

* Younger than 10 years or older than 17 years.
* No IBD diagnosis, or IBD diagnosed less than 6 months ago.
* Associated chronic condition (neurological, metabolic, psychiatric, or other) likely to interfere with questionnaire completion or interview participation.
* Major language or cognitive impairment preventing adequate understanding or interview participation.
* Not affiliated to, or not beneficiary of, a social security scheme.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Aged 10 to 17 years at inclusion.
  * Diagnosed inflammatory bowel disease (Crohn's disease or ulcerative colitis) confirmed and diagnosed for at least 6 months.
  * Followed in the pediatric gastroenterology department at Hôpital Lenval (CHU de Nice).
  * Sufficient cognitive and language abilities to understand questionnaires and participate in an individual interview.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Perceived barriers and facilitators to regular physical activity | at the inclusion
  Assessed through a single semi-structured interview. Qualitative thematic analysis will be used to identify and categorize perceived barriers and facilitators to regular physical activity in pediatric IBD.

SECONDARY OUTCOMES:
Physical activity level and sedentary behavior (CAPAS-Q) | at the inclusion
  Measured using the CAPAS-Q self-administered questionnaire to describe participants' physical activity and sedentary behavior.
Health-related quality of life (IMPACT-III) | at the inclusion
  Measured using the IMPACT-III self-administered questionnaire to assess health-related quality of life in pediatric IBD.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Lenval Hôpitaux pédiatrique Nice CHU Lenval, Nice, France

IPD SHARING:
Plan to Share IPD: No